CLINICAL TRIAL: NCT04621578
Title: The Effect of Prevention and Treatment of Transcutaneous Electrical Acupoint Stimulation on Postoperative Dizziness in Patients With Hemifacial Spasm Undergoing Microvascular Decompression Surgery: A Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation on Postoperative Dizziness in Hemifacial Spasm Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chief of the Anesthesiology Department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020PHB232-01
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Transcutaneous Electrical Acupoint Stimulation; Hemifacial Spasm; Dizziness
MeSH Terms: conditions — Hemifacial Spasm; Dizziness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical acupoint stimulation arm (Experimental): Patients will be given TEAS treatment at the maximum tolerable intensity at a frequency of 2 Hertz (Hz) after surgery in postanesthesia care unit (PACU), and after returning to the ward.
  Interventions: Device: HANS 100B stimulator (4 conductors, 8 electrodes; Jisheng Co., Nanjing, China)
- Sham stimulation arm (Sham Comparator): Patients will use the same device, same stimulation site, and be treated at the same time points, but the lead of the device was damaged. Therefore, although the patients can see the stimulator running, there is actually no current passing through.
  Interventions: Device: HANS 100B stimulator (4 conductors, 8 electrodes; Jisheng Co., Nanjing, China)

INTERVENTIONS:
Device: HANS 100B stimulator (4 conductors, 8 electrodes; Jisheng Co., Nanjing, China) — Stimulation sites: Mastoid area on the contralateral side of the operation, Fengchi acupoint on the contralateral side of the operation, and Neiguan acupoints on both sides.
  Timing of stimulation: In postanesthesia care unit (PACU) after extubation, 6 hours, 24 hours, 48 hours, and 72 hours after returning to the ward. 30-minutes treatment for each time-point.

SUMMARY:
To observe the prevention and treatment effect of transcutaneous electrical acupoint stimulation (TEAS) on postoperative dizziness in patients with hemifacial spasm undergoing microvascular decompression surgery, and its possible mechanisms.

DETAILED DESCRIPTION:
Hemifacial spasm (HFS) is mainly caused by vascular compression on the roots of the VII cranial nerves from the brain stem. Microvascular decompression (MVD) is the exact surgical method for the treatment of HFS, but the incidence of dizziness and postoperative nausea and vomiting (PONV) after MVD is extremely high. Despite the use of dual antiemetic therapy during the operation, the incidence of PONV within 24 hours after MVD is still as high as 66.7%. Medication alone has limited effects on dizziness and PONV treatment after MVD. Meta-analysis shows that transcutaneous electrical acupoint stimulation (TEAS) is associated with the reduction of post-emetic remedies and the incidence of dizziness after general anesthesia, and it can be integrated into the multi-modal therapy of PONV. Therefore, the purpose of our study is to observe the prevention and treatment effect of TEAS on postoperative dizziness in patients with hemifacial spasm undergoing microvascular decompression surgery, and explore its possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status: I-III
* Body mass index (BMI): 18-30
* Diagnosed of hemifacial spasm
* Undergoing microvascular decompression surgery

Exclusion Criteria:

* Pregnant or lactating women
* Poorly controlled hypertension or poorly controlled diabetes, severe cardiovascular and cerebrovascular diseases and mental illness
* Cardiac pacemakers
* Scars on bilateral Neiguan acupoints or on the mastoid area
* Upper limb nerve injury
* Raynaud's syndrome
* Motion sickness or PONV history
* Eye diseases (glaucoma, cataracts, eye trauma, etc.) or previous eye surgery
* Participate in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
The incidence of dizziness at 2 hours after returning to the ward on the day of surgery | 2 hours after returning to the ward on the day of surgery
  The patients and their families will be asked to record a diary about their symptoms of dizziness, nausea, vomiting and headache after surgery, and they will be followed up after surgery.

SECONDARY OUTCOMES:
Numerical rating scale (NRS) score of postoperative dizziness | In PACU after extubation, and 2 hours, 6 hours, 24 hours, 48 hours, 72 hours after returning to the ward.
  A 0-10 point numerical rating scale (NRS) will be used for evaluation of the severity of postoperative dizziness. 0 means no dizziness, and 10 means very severe dizziness. The degree of dizziness worsens as the number increases.
The incidence and severity of postoperative nausea | In PACU after extubation, and 2 hours, 6 hours, 24 hours, 48 hours, 72 hours after returning to the ward.
  Nausea severity will be evaluated by a 0-10 point numerical rating scale (NRS). 0 means no nausea, and 10 means very severe nausea. The degree of nausea worsens as the number increases.
The number of vomiting after surgery | In PACU after extubation, and 2 hours, 6 hours, 24 hours, 48 hours, 72 hours after returning to the ward.
  Vomiting times after surgery.
The use of remedial drugs after surgery | From the day of surgery to 72 hours after surgery.
  Drug used for anti-emetic or anti-dizziness after surgery.
The incidence and severity of postoperative headache | In PACU after extubation, and 2 hours, 6 hours, 24 hours, 48 hours, 72 hours after returning to the ward.
  Headache severity will be evaluated by a 0-10 point numerical rating scale (NRS). 0 means no headache, and 10 means very severe headache. The degree of headache worsens as the number increases.
Changes in intraocular pressure before and after surgery | Before anesthesia induction, and before leaving PACU on the day of surgery.
  Intraocular pressure will be measured by a non-contact tonometer before and after surgery by the same operator.
Gastrin and 5-Hydroxytryptamine (5-HT) levels in serum and cerebrospinal fluid | The peripheral blood samples will be collected on the day of surgery, and on postoperative day 1. The CSF samples will be collected on the day of surgery.
  Peripheral blood will be collected before and after surgery, and cerebrospinal fluid (CSF) will be collected during the surgery.
Postoperative complications monitoring | From the day of surgery to the day of discharge.
  The Clavien-Dindo grading system will be used.
Postoperative duration of stay in hospital | From the day of surgery to the day of discharge.
  The duration when patients stay in hospital after surgery.
Dizziness symptoms 4 weeks after discharge | 4 weeks after discharge.
  Patients will be followed up by telephone 4 weeks after discharge, and the Dizziness Handicap Inventory (DHI) will be used for measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Miller LE, Miller VM. Safety and effectiveness of microvascular decompression for treatment of hemifacial spasm: a systematic review. Br J Neurosurg. 2012 Aug;26(4):438-44. doi: 10.3109/02688697.2011.641613. Epub 2011 Dec 15. PMID 22168965
- [Background] Thongrong C, Chullabodhi P, Kasemsiri P, Kitkhuandee A, Plailaharn N, Sabangban L, Jimarsa T. Effects of Intraoperative Dexamethasone and Ondansetron on Postoperative Nausea and Vomiting in Microvascular Decompression Surgery: A Randomized Controlled Study. Anesthesiol Res Pract. 2018 Nov 11;2018:6297362. doi: 10.1155/2018/6297362. eCollection 2018. PMID 30534153
- [Background] Chen J, Tu Q, Miao S, Zhou Z, Hu S. Transcutaneous electrical acupoint stimulation for preventing postoperative nausea and vomiting after general anesthesia: A meta-analysis of randomized controlled trials. Int J Surg. 2020 Jan;73:57-64. doi: 10.1016/j.ijsu.2019.10.036. Epub 2019 Nov 6. PMID 31704425